CLINICAL TRIAL: NCT02915380
Title: Pituitary Dysfunction After Aneurysmal Subarachnoid Hemorrhage
Acronym: TIRASH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Rita Bertuetti (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Dr. Rita Bertuetti, Medical Doctor, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: TIRASH-1.0
Record Dates: First submitted 2016-09-06; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Thyroid Disfunction; Subarachnoid Haemorrhage From Cerebral Aneurism Rupture; Pituitary Disfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Evaluation of pituitary endocrine function — The basal thyroid hormone and test to perform will be: TSH, fT4, fT3.
  When available, the following hormones will be tested:
  FSH, LH, estradiol (in women), testosterone (in men), sex hormone-binding globulin (SHBG), ACTH, cortisol, prolactin, Na, K; serum levels of GH and IGF-1; and serum and urine osmolality.
  Adrenal function will be evaluated through ACTH-stimulation testing . Adrenal or GH insufficiency will be evaluated by insulin tolerance testing (ITT)
Behavioral: Evaluation of clinical outcome — Patients' outcome will be assessed as modified Rankin Scale (mRS) at discharge from the hospital, at 3, 6 and 12 months.
Behavioral: Evaluation of neuropsychological function — Neuropsychological examination will be conducted focusing on verbal comprehension (Token Test) and visual neglect. Verbal and visual short term and working memory visuospatial construction and figural memory will be performed through Rey Osterrieth Complex figure test, and psychomotor speed attention and concentration through Trail Making Test.

SUMMARY:
Recently, the occurrence and potential impact of pituitary dysfunction after aSAH has gained increasing interest. Several studies have demonstrated pituitary dysfunction after SAH suggesting that pituitary dysfunction may be a contributing factor for residual symptoms after SAH. This is an observational multicentric study aimed to test the prevalence of thyroid abnormalities, other neuroendocrinological dysfunction and their influence on outcome of patients affected by aSAH.

DETAILED DESCRIPTION:
The incidence of aneurysmal subarachnoid hemorrhage (aSAH) varies between 6 to 10/100,000 subjects per year and it is a major cause of death and disability. The mortality rate ranges from 40 to 50%, and those who do survive SAH have high rates of functional limitations that could lead to impaired quality of life, including fatigue, depression, and loss of motivation.

Because aSAH affects patients in their most productive years of life, the disease has important social, and economic implications, and early prediction of long-term outcome is based on multiple factors including the primary injury secondary insults as well as neurorehabilitation interventions.

Recently, the occurrence and potential impact of pituitary dysfunction after aSAH has gained increasing interest. Several studies have demonstrated pituitary dysfunction after SAH suggesting that pituitary dysfunction may be a contributing factor for residual symptoms after SAH. However, questions remain about the real prevalence and impact of such dysfunction on patients' outcome both in the acute and chronic phase after these events.

In two recent metanalysis, the prevalence of total pituitary dysfunction was found with pooled frequencies of 0.31 (95% confidence interval CI: 0.22-0.43) [Can et a.] and 49.3.0% (95% CI 41.6%-56.9%) [Robba et al] during the acute phase (< 6 months from aSAH) and decreasing in the chronic phase to 0.25 (95% CI: 0.16-0.36) [Can et al.] and 25.6% (95% CI 18.0%-35.1%) [Robba et al]. However, the authors found high heterogenicity and different results between the available literature; many differences were found in the in the choice of time of pituitary function assessment and SAH, of diagnostic criteria and units of measurement used to establish the diagnosis of hypopituitarism after SAH.

Finally, it is not clear which is the hormone axis more likely to be affected after aSAH.

It is believed that, among the other, the incidence of thyroid dysfunction is the most relevant, as it is associated with severe clinical impairment and symptoms. In literature, the prevalence of thyroid dysfunction after aSAH is reported from 0 to 35%.[Karaka, Tanrivedi].

Hypothyroidism includes a wide variety of symptoms including weakness, fatigue, depression, irritability, memory loss and decreased libido. Should these abnormalities complicate more than one third of the patients, hormone testing and eventually replacement should become "standard of care" to test.

In order to define the actual incidence of these abnormalities, an observational multicentric study to test thyroid abnormalities, including TSH, fT4 (free thyroxine) and fT3 (free triiodothyronine) changes, is warranted.

Secondary endpoints of such study include the prevalence of other neuroendocrinological dysfunction and their influence on the patients' outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute aneurysmal SAH aged between 18 and 70 years of age who could be subjected to endocrine evaluation within 10 days of ictus and at follow-up.

Exclusion Criteria:

* be major depression, psychiatric premorbidity, pituitary adenoma or perisellar lesion,preexisting hypopituitarism of any degree, previous hormonal substitution, patients in moribund state, pregnancy, glucocorticoid medication on admission to hospital or during treatment, prior pituitary insufficiency, and unsalvageable aSAH.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for aneurysmal subarachnoid haemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of thyroid disfunction | At 2 weeks after aSAH
  Thyroid-stimulating hormone (TSH), free thyroxin (fT4), free triiodothyronine (fT3).
Incidence of thyroid disfunction | 3 months after aSAH
  Thyroid-stimulating hormone (TSH), free thyroxin (fT4), free triiodothyronine (fT3).
Incidence of thyroid disfunction | 6 months after aSAH
  Thyroid-stimulating hormone (TSH), free thyroxin (fT4), free triiodothyronine (fT3).
Incidence of thyroid disfunction | 12 months after aSAH
  Thyroid-stimulating hormone (TSH), free thyroxin (fT4), free triiodothyronine (fT3).

SECONDARY OUTCOMES:
Incidence of pituitary- sexual hormones disfunction | At 2 weeks, and at follow up at 3, 6 and 12 months.
  serum levels of follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol (in women), testosterone (in men), sex hormone-binding globulin (SHBG).
Survival | At 2 weeks, and at follow up at 3, 6 and 12 months
  Modified Ranking Scale
Incidence of pituitary-adrenal axis disfunction | At 2 weeks, and at follow up at 3, 6 and 12 months.
  Serum levels of adrenocortico-tropic hormone (ACTH), cortisol, Na, K; serum and urine osmolality. Adrenal function will be evaluated through ACTH-stimulation testing with injection of 250 mcg of ACTH, and a peak of cortisol <500 nmol/l will be considered pathologic. Adrenal or GH insufficiency will be evaluated by insulin tolerance testing (ITT), and peak response of more than 3ng/ml for GH and and 500 nmol/l for cortisol will be considered as normal.
Incidence of growth hormone insufficiency | At 2 weeks, and at follow up at 3, 6 and 12 months
  serum levels of growth hormone (GH) and insulin-like growth factor 1 (IGF-1). Adrenal or GH insufficiency will be evaluated by insulin tolerance testing (ITT), and peak response of more than 3ng/ml for GH and and 500 nmol/l for cortisol will be considered as normal.
Incidence of language disorders | At 2 weeks, and at follow up at 3, 6 and 12 months
  Neuropsychological examination focused on verbal comprehension will be evaluated through the application of Token Test .
  Incidence of impaired scoring will be correlated to incidence of altered hormone levels detected in the blood.
Incidence of memory disorders | At 2 weeks, and at follow up at 3, 6 and 12 months
  Verbal and visual short term and working memory visuospatial construction and figural memory will be performed through Rey Osterrieth Complex figure test.
  Incidence of impaired scoring will be correlated to incidence of altered hormone levels detected in the blood.
Incidence of attention disorders | At 2 weeks, and at follow up at 3, 6 and 12 months
  Psychomotor speed attention and concentration will be assessed through Trail Making Test.
  Incidence of impaired scoring will be correlated to incidence of altered hormone levels detected in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Robba, MD, Study Director — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided